CLINICAL TRIAL: NCT01300286
Title: Open Label Use Of RiaStap During Aortic Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024305
Record Dates: First submitted 2011-01-09; First posted 2011-02-21 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-01

CONDITIONS: Coagulopathic Bleeding
MeSH Terms: interventions — Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RiaSTAP (Experimental): One time dose of 70 mg/kg will be administered intravenously.
  Interventions: Drug: RiaSTAP

INTERVENTIONS:
Drug: RiaSTAP — One time dose of 70 mg/kg will be administered intravenously.

SUMMARY:
The overall purpose of this study is to administer fibrinogen concentrate (RiaSTAP, CSL Behring, Marburg, Germany) with the goal of treating coagulopathic bleeding by improving hemostasis thereby reducing overall blood product transfusion after separation from cardiopulmonary bypass following aortic reconstructive surgery. With the current sample size this is a pilot study and in effect will determine the fibrinogen level response to fibrinogen concentrate administered during aortic reconstructive surgery. It will be underpowered to detect reduction in bleeding but comparison to historical controls will be included as a secondary outcome.

DETAILED DESCRIPTION:
Study design Open-label study Inclusion criteria Elective, adult aortic reconstruction involving a hemi-arch replacement at Duke University Medical Center (DUMC).

Exclusion criteria Concomitant procedures such as Coronary Artery Bypass Grafting (CABG) , stents (within the last 3 years), refusal of blood transfusion, recent Myocardial Infarction (MI) (within the last 3 months), pregnancy, INR > 1.1, platelet inhibitor drugs within 5 days of surgery (aspirin 325 mg within 48 hours of surgery), platelet count < 150,000, age <18 years, inability to obtain written informed consent, known coagulopathy including a history of recent coumadin therapy.

Primary outcome variable Fibrinogen level Secondary outcome variables Total blood product units administered during post op day (POD) 0, 1, 2, 12 and 24 hour chest tube drainage, ventilator time, duration of oxygen dependency, renal dysfunction. Adverse events will be recorded.

Study procedure The administration of RiaSTAP is detailed in the flowchart below.

Projected milestones Based on recent surgical volume and assuming a conservative recruitment in the 60-70% range we will plan to complete the study of 22 patients as determined by budgetary constraints in a projected 12-month study period.

We plan to evaluate the protocol after 11 (half of the) patients. Reevaluation and modification may include broadening the inclusion criteria and/or altering our transfusion protocol depending on the results of the first 11 patients and the projected recruitment rate.

Safety monitoring Adverse events as recorded in the aortic database of historical controls will form the basis of the clinical research form (CRF) and are specifically outlined and defined below.

The conduct of anesthesia and surgery will be at the discretion of the attending surgeon and anesthesiologist. Following heparin reversal with protamine sulphate and administration of 30mcg/kg DDAVP and 5g aminocaproic acid as per standard practice for these cases, surgical hemorrhage will be excluded by the attending surgeon. The dose of fibrinogen concentrate will be administered as described in the Figure. RiaSTAP will only be administered if coagulopathic bleeding is observed by the surgeon such that it will be used for the treatment, not the prevention of bleeding.

It is standard practice for the surgeon to report coagulopathic bleeding (as defined by lack of visible clot in the wound, soaking of swabs with blood and/or continued aspiration of blood into the cell-saver device) before we administer blood products and/or rFVIIa after separation from bypass and following administration of protamine to reverse heparin, aminocaproic acid to inhibit fibrinolysis and DDAVP to augment platelet function.

The Food and Drug (FDA) approved dose of 70mg/kg will be used. Following the dosage of fibrinogen concentrate subsequent care of the patient will not be governed by the study protocol. Specifically, transfusion of blood products are suggested in the flow diagram above and transfusion guidelines have been developed by Dr Ian Welsby and Dr Chad Hughes in August 2009 in response to difficulties managing such cases and both of these will be available for use, BUT will only be applied at the discretion of the attending anesthesiologist and surgeon.

Proposed laboratory tests in addition to standard of care Time points

1. Baseline Anesthesia induction
2. Pre RiaSTAP After separation from cardio pulmonary bypass (CPB), after desired protamine given
3. Post RiaSTAP Ten minutes after RiaSTAP administered
4. Post op On admission to intensive care unit (ICU)
5. Post op 24 hours after surgery Plasma Heparin level (to avoid misinterpretation of clot based factor assays) Thrombin clot time (as above) Fibrinogen (Clauss method) Clotting Factor Levels Endogenous thrombin potential Whole blood Rotational Thromboelastometry (ROTEM) including Fibrinogen Test (FIBTEM) but not Lysis Test (APTEM) MEA platelet aggregometry (to be provided by CSL Behring)

20ml of blood will be drawn at each timepoint, total 100ml.

ELIGIBILITY:
Inclusion Criteria:

* Elective, adult aortic reconstruction involving a hemi-arch replacement at DUMC.

Exclusion Criteria:

* Concomitant procedures such as CABG , stents (within the last 3 years), refusal of blood transfusion, recent MI (within the last 3 months), pregnancy, INR > 1.1, platelet inhibitor drugs within 5 days of surgery (aspirin 325 mg within 48 hours of surgery), platelet count < 150,000, age <18 years, inability to obtain written informed consent, known coagulopathy including a history of recent coumadin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Welsby, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Rahe-Meyer N, Pichlmaier M, Haverich A, Solomon C, Winterhalter M, Piepenbrock S, Tanaka KA. Bleeding management with fibrinogen concentrate targeting a high-normal plasma fibrinogen level: a pilot study. Br J Anaesth. 2009 Jun;102(6):785-92. doi: 10.1093/bja/aep089. Epub 2009 May 2. PMID 19411671
- [Background] Peyvandi F, Haertel S, Knaub S, Mannucci PM. Incidence of bleeding symptoms in 100 patients with inherited afibrinogenemia or hypofibrinogenemia. J Thromb Haemost. 2006 Jul;4(7):1634-7. doi: 10.1111/j.1538-7836.2006.02014.x. No abstract available. PMID 16839371
- [Background] Rahe-Meyer N, Solomon C, Winterhalter M, Piepenbrock S, Tanaka K, Haverich A, Pichlmaier M. Thromboelastometry-guided administration of fibrinogen concentrate for the treatment of excessive intraoperative bleeding in thoracoabdominal aortic aneurysm surgery. J Thorac Cardiovasc Surg. 2009 Sep;138(3):694-702. doi: 10.1016/j.jtcvs.2008.11.065. Epub 2009 May 17. PMID 19698858
- [Background] Kreuz W et al Tranfus Apheresis Sci 2005; 32: 239-46
- [Background] Lind P, Hedblad B, Stavenow L, Janzon L, Eriksson KF, Lindgarde F. Influence of plasma fibrinogen levels on the incidence of myocardial infarction and death is modified by other inflammation-sensitive proteins: a long-term cohort study. Arterioscler Thromb Vasc Biol. 2001 Mar;21(3):452-8. doi: 10.1161/01.atv.21.3.452. PMID 11231928

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RiaSTAP
Started | 23
Completed | 22
Not Completed | 1
Not completed — did not get dosed | 1

BASELINE CHARACTERISTICS:
Arm/Group | RiaSTAP
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Fibrinogen Level Change
Description: Fibrinogen levels will be assessed only at the timepoints listed in the timeframe and for a maximum of 24 hours.
Time Frame: Anesthesia Induction (Baseline), Pre RiaSTAP (est. 4 hr after baseline), Post RiaSTAP (est: 10 minutes after RiaSTAP administered), ICU Admission (est. 6 hours after baseline), 24 Hour post op (est: 24-30 hr after baseline)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | RiaSTAP
Number analyzed (Participants) | 22
mg/dl
  Anesthesia Induction,I | 317 (49)
  Pre RiaSTAP | 235 (39)
  Post RiaSTAP | 331 (41)
  ICU admission | 312 (41)
  24 hours post op | 372 (45)

2. Secondary Outcome: Packed Red Blood Cell Transfusion
Time Frame: Anesthesia Induction (Baseline), after CPB, ICU Admission (est. 6 hours after baseline) to post op day 2 (est: 30- 54 hr after baseline)
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | RiaSTAP
Number analyzed (Participants) | 22
units | 1 [0 to 2]

3. Secondary Outcome: Fresh Frozen Plasma Transfusion
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | RiaSTAP
Number analyzed (Participants) | 22
mL | 1000 [1000 to 1500]

4. Secondary Outcome: Platelet Transfusion
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | RiaSTAP
Number analyzed (Participants) | 22
mL | 400 [274 to 592]

5. Secondary Outcome: Cryoprecipitate Transfusion
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | RiaSTAP
Number analyzed (Participants) | 22
mL | 20 (59)

ADVERSE EVENTS:
Arm/Group | RiaSTAP
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 6/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RiaSTAP (N=22)
Postoperative atrial fibrillation (Cardiac disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No